CLINICAL TRIAL: NCT03013075
Title: Comparative Effect of Combined High Spinal and General Anaesthesia With General Anaesthesia Alone On Right Ventricular Function In Patients With Mitral Valvular Disease With Pulmonary Hypertension
Brief Title: General Plus Spinal Anesthesia and General Anesthesia Alone on Right Ventricular Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ganesh Kumar Munirathinam, Fellow resident, Department of anesthesia and intensive care, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INT/IEC/2016/2573
Record Dates: First submitted 2017-01-02; First posted 2017-01-06 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Anesthesia, Spinal; Morphine; Anesthetics, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPINAL PLUS GENERAL ANESTHESIA (Experimental): Patient will receive the intervention SPINAL ANESTHESIA before the start of surgery using Bupivacaine heavy 40 mg and Morphine 250 micro grams comprising a total volume of 8 ml to achieve a spinal block up to T2 level followed by general anesthesia
  Interventions: Procedure: Spinal anesthesia with Bupivacaine heavy and Morphine; Drug: Bupivacaine heavy and Morphine; Drug: General Anesthetics
- ONLY GENERAL ANESTHESIA (Active Comparator): Patient will receive only general anesthesia before the start of surgery
  Interventions: Drug: General Anesthetics

INTERVENTIONS:
Procedure: Spinal anesthesia with Bupivacaine heavy and Morphine — Spinal anesthesia with Bupivacaine heavy 40 mg and Morphine 250 micro grams will be given to patient in addition to the routine general anesthesia before the start of surgery
  Arms: SPINAL PLUS GENERAL ANESTHESIA
Drug: Bupivacaine heavy and Morphine
  Arms: SPINAL PLUS GENERAL ANESTHESIA
Drug: General Anesthetics

SUMMARY:
The investigator hypothesize that High Spinal Anesthesia (HSA) by its effect on attenuation of stress response, decrease in pulmonary vascular resistance, myocardial protection and positive myocardial oxygen balance will cause improvement in right ventricular function. So far there is no study that has evaluated the effect of HSA anesthesia on the right ventricular function, hence the investigator planned this study to compare the effect of HSA on the right ventricular function in patients with mitral valve disease with moderate to severe pulmonary hypertension planned for mitral valve replacement surgery.

DETAILED DESCRIPTION:
All study patients will undergo routine TTE and TEE examination protocol followed at the investigator institution. All the other routine monitoring such as end tidal carbon dioxide, urine output, ABG, ACT, BIS, electrolytes, blood sugar, hemoglobin and ventilatory parameters etc for open heart surgery will be done as per institutional practice. In the study group, the patients will receive spinal anesthesia after placement of invasive lines and prior to induction of GA.In both the study group GA will be induced with midazolam 1-2 mg, fentanyl 2μ/kg and propofol titrated to achieve loss of consciousness. Inj. Vecuronium bromide 0.1mg/kg will be used as muscle relaxant to facilitate tracheal intubation and lignocaine spray (LOX 10% spray, Neon laboratories LTD, Thane, India) will be used over vocal cords prior to intubation to blunt the sympathetic stimulation.

Subsequently anesthesia will be maintained in both the groups, with isoflurane inhalation to maintain BIS values between 40 to 60. In control group, fentanyl infusion 1μ/kg/hr will be started for analgesia, a similar looking infusion without fentanyl will be started in the spinal group.All patients will be shifted to ICU with inotropic and vasopressor support as per the hemodynamic condition.

ELIGIBILITY:
Inclusion Criteria:

* 50 consecutive patients of 18 to 60 years age,
* NYHA class II or III,
* with mitral valvular disease with moderate to severe PAH (mean pulmonary artery pressure > 40 mmHg) undergoing MVR

Exclusion Criteria:

* emergency or redo surgery, patients with associated CAD or other valvular heart disease,
* COPD,
* bronchial asthma,
* obesity (BMI more than 30), anticipated difficult airway,
* opioid drug abuse or addiction and those with contraindication for spinal anaesthesia including local site infection,
* spinal deformity, deranged coagulogram defined by platelet count < 80,000 & INR > 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of right ventricular function defined by 20% increase in the TAPSE in the study group when compared to the control group | Till patient got discharged from ICU, an average of 5 days

SECONDARY OUTCOMES:
Pulmonary vascular resistance | Till patient got discharged from ICU, an average of 5 days
Left ventricular ejection fraction | Till patient got discharged from ICU, an average of 5 days
Right ventricular myocardial performance index | Till patient got discharged from ICU, an average of 5 days
Mechanical ventilation duration | Till patient got discharged from ICU, an average of 5 days
Intensive care unit stay | Till patient got discharged from ICU, an average of 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India